CLINICAL TRIAL: NCT00627120
Title: A Placebo-Controlled, Ascending Single-Dose Study to Evaluate the Safety and Pharmacokinetics of VGX-1027 in Healthy Subjects
Brief Title: Phase I Safety and Pharmacokinetic Study of VGX-1027 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VGX Pharmaceuticals, LLC (Industry)
Collaborators: GeneOne Life Science, Inc. (Industry)
Responsible Party: C. Jo White, MD, VGX Pharmaceuticals, Inc
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CAT001
Record Dates: First submitted 2008-01-17; First posted 2008-02-29 (Estimated); Last update posted 2009-01-09 (Estimated); Status verified 2009-01

CONDITIONS: Healthy
Keywords: healthy volunteers
MeSH Terms: interventions — 3-phenyl-4,5-dihydro-5-isoxazole acetic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental): 1mg dose group
  Interventions: Drug: VGX-1027
- 2 (Experimental): 10mg dose group
  Interventions: Drug: VGX-1027
- 3 (Experimental): 100mg dose group
  Interventions: Drug: VGX-1027
- 4 (Experimental): 200mg dose group
  Interventions: Drug: VGX-1027
- 5 (Experimental): 400mg dose group
  Interventions: Drug: VGX-1027
- 6 (Experimental): 800mg dose group
  Interventions: Drug: VGX-1027

INTERVENTIONS:
Drug: VGX-1027 — Subject will be given a single dose of VGX-1027 ranging from 1-800mg and monitored for safety and pharmacokinetics for 8 days.

SUMMARY:
To assess the safety and tolerability of a single dose of VGX-1027 in the range of 1-800mg.

DETAILED DESCRIPTION:
This study will evaluate:

* The safety and tolerability of a single dose of VGX-1027 as determined by: adverse event reporting, clinical laboratory results, vital signs, physical examinations, and electrocardiograms (ECGs).
* The pharmacokinetic (PK) profile of VGX-1027 maximum concentration (Cmax)

ELIGIBILITY:
Inclusion Criteria:

* Must give written informed consent.
* Healthy subjects as determined by no clinically significant deviation from normal as judged by the investigator in medical history, physical examination, ECGs and clinical laboratory evaluations
* Body Mass Index of 18-30kg/m^2 inclusive
* Males or females ages 18-60, inclusive. Women who are not of childbearing potential may enroll. Women must have a negative pregnancy test within 72 hours prior to start of study drug administration or be surgically sterile.

Exclusion Criteria:

* Women who are of childbearing potential
* Women who are pregnant or breastfeeding
* Women with a positive pregnancy test on enrollment or prior to study drug administration
* Male subjects who are unwilling to agree to practice barrier contraception during the study and for three months following dosing
* Any significant acute or chronic mental illness
* Current or recent gastrointestinal disease that may impact the absorption of the drug
* Any major surgery within 4 weeks of enrollment
* Donation of blood or plasma to a blood bank or in a clinical study (except screening visit) within 4 weeks of enrollment
* Blood transfusion within 4 weeks of enrollment
* Inability to tolerate oral medication
* Inability to be venipunctured and/or tolerate venous access
* Recent (within 6 months) drug or alcohol abuse
* History of bleeding disorder
* History of head trauma or seizures
* Any other sound medical, psychiatric and/or social reason as determined by the Investigator
* Evidence of organ dysfunction or any clinically significant deviation from normal in vital signs, physical examination, ECG, or clinical laboratory determinations
* Positive urine screen for drugs of abuse
* Positive blood screen for hepatitis C antibody, hepatitis B surface antigen, HIV 1/2 antibody
* History of any significant drug allergy
* Exposure to any investigational drug within 4 weeks prior to enrollment or greater that 4 weeks for investigational drugs that may have a longer half-life
* Use of any prescription drugs or over the counter acid controllers within 4 weeks prior to enrollment
* Use of any other drugs, including over the counter vitamins, medications and/or herbal preparations within 2 weeks prior to enrollment
* Use of oral, injectable or implantable hormonal contraceptive agents within 3 months prior to enrollment
* Use of alcohol containing beverages within 1 week prior to enrollment
* Use of grapefruit containing products within 1 week prior to enrollment
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g. infectious disease) illness must not be enrolled into this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Safety as determined by vital signs, physical examinations, ECGs, clinical laboratory evaluations, and AE reporting. | Day 8

SECONDARY OUTCOMES:
Pharmacokinetics | Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Stephan A Bart, MD, Principal Investigator — SNBL Clinical Pharmacology Center, Inc.
Locations (1):
- SNBL Clinical Pharmacology Center, Baltimore, Maryland, United States